CLINICAL TRIAL: NCT04620239
Title: Multicenter Phase 3 Pivotal Study to Evaluate the Safety and Efficacy of TOOKAD (Padeliporfin) Vascular Targeted Photodynamic Therapy in the Treatment of Low Grade Upper Tract Urothelial Cancer
Brief Title: ENdoluminal LIGHT ActivatED Treatment of Upper Tract Urothelial Cancer (ENLIGHTED) Study
Acronym: UCM301
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Steba Biotech S.A. (Other)
Collaborators: PrimeVigilance (Industry); ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN2001 UCM301
Record Dates: First submitted 2020-11-05; First posted 2020-11-06 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Transitional Cell Cancer of Renal Pelvis and Ureter
Keywords: UTUC; Low Grade
MeSH Terms: interventions — padeliporfin

STUDY DESIGN:
Intervention Model Description: Phase III, single arm, non randomized, multicenter trial
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- padeliporfin VTP (Experimental): Induction Treatment phase:1-3 padeliporfin VTP treatments provided 4 weeks (28 +/-3 days) apart.
  Maintenance Treatment Phase: Repeated maintenance VTP treatments during this period will be provided for patients who show evidence of tumor recurrence that is deemed treatable.
  Interventions: Drug: padeliporfin VTP

INTERVENTIONS:
Drug: padeliporfin VTP — During treatment, placement at the target area of an optical light fiber, through the working channel of the ureteroscope. Intravenous administration of padeliporfin at the dose of 3.66 mg/kg infused over 10 minutes. Each target area will be illuminated for 10 minutes.
  Other Names: WST11

SUMMARY:
This is a phase 3, open label, single arm study of padeliporfin in the treatment of Upper Tract Urothelial Carcinoma (UTUC). The ENLIGHTED study will recruit patients with low-grade non-invasive upper tract urothelial carcinoma in either the kidney or the ureter. Patients will be treated with padeliporfin VTP in two phases: an Induction Treatment Phase and a Maintenance Treatment Phase and will be followed up for up to an additional 48 months in the long term (non intervention) follow up phase with the specific duration depending on the patient's response to treatment

DETAILED DESCRIPTION:
Induction Treament Phase: Patients entered in the study will undergo an induction treatment phase consisting of 1-3 padeliporfin VTP treatments provided 4 weeks (28 +/-3 days) apart. The goal of this induction treatment phase will be to achieve Complete Response (CR) in the involved ipsilateral tract system. During this phase, patients will be treated with padeliporfin VTP to visually identified tumor sites in the calyces, renal pelvis and/or ureter and subsequently examined endoscopically at 28 +/- 3 days post treatment to determine whether the treatment was successful. If CR is not achieved, an additional two treatments of padeliporfin VTP are permitted 28 +/- 3 days apart for a total of up to 3 treatments during the induction treatment phase. The Primary Response Evaluation (PRE) will be performed 28 +/- 3 days after the last VTP treatment, to determine if the treatment was successful at achieving CR defined as: absence of visible tumor on endoscopy, negative urinary cytology by instrumented collection, and no evidence of tumor on biopsy (if feasible). Patients undergoing extirpative surgery of any part of the ipsilateral kidney or ureter for indications related to urothelial cancer will be considered as no longer having CR. If CR is not achieved after 3 treatments with padeliporfin VTP the treatment will be considered unsuccessful and the patient will be discontinued from the Treatment Phases.

Maintenance Treatment Phase: Patients achieving CR at the induction treatment phase will be allowed into the maintenance treatment phase of the study. The patients will then be followed over a period of 12 months post PRE, to assess the duration of response and its safety, and to provide planned maintenance treatment.

Repeated maintenance VTP treatments during this period will be provided for patients who show evidence of tumor recurrence that is deemed treatable as defined by the following criteria: low-grade tumors with the largest tumor (index tumor) betwen 5 mm and 15 mm in diameter, in up to 2 anatomical locations in the calyces, renal pelvis or the ureter with ureter involvement in one anatomical location with no more than 20 mm of contiguous ureteral length). Patients with treatable tumor recurrence post Induction Treatment Phase would be considered as no longer having 'complete response in the entire ipsilateral kidney' and time to recurrence will be recorded. Patients undergoing extirpative surgery of any part of the ipsilateral kidney or ureter for indications related to urothelial cancer will be considered as no longer having CR and time to this event will be recorded.

Long Term Follow-up Phase: Patients completing the 12 months of the maintenance treatment phase of the study, could be followed for an additional 48 months to monitor for disease related outcomes and VTP treatment related adverse events with the specific duration depending on the patient's response to treatment. No additional padeliporfin VTP treatment will be administered during this phase. Patients completing the maintenance phase of the study who are in CR in V3 will undergo additional assessments 18 and 24 months (+/- 1 month) post-PRE and annually thereafter and for up to 5 years post PRE or until recurrence, progression, death or loss to follow up, to document safety and ongoing response.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 years or older
* Able to understand and provide written informed consent and willing to comply with all tests and procedures associated with the study
* New or recurrent low-grade, non-invasive UTUC disease
* Biopsy-proven disease . A concurrence of the central pathology reader will be required for eligibility.
* Up to 2 biopsy-proven sites of low-grade involvement with the largest tumor (index tumor) between 5 mm and 15 mm in diameter (as measured by endoscopy), both located in the calyces,renal pelvis or in the ureter of the ipsilateral kidney, with an absence of high-grade cells on cytology. (Ureter involvement should be in one anatomical location with no more than 20 mm of contiguous ureteral length)
* Karnofsky Performance Status ≥ 50%
* Adequate organ function defined at baseline as:

  * ANC ≥1,000/ μl,
  * Platelets ≥75,000/ μl, Hb ≥9 g/dl,
  * INR ≤ 2
  * Estimated glomerular giltration rate (eGFR) ≥30 ml/min (using CKD-EPI Method)
  * Total serum bilirubin <3 mg/dL, AST/ALT ≤5× upper limit of normal

Exclusion Criteria:

* Current high-grade or muscle invasive (>pT1) urothelial carcinoma of the bladder
* Carcinoma in situ (CIS) current or previous in the upper urinary tract
* History of invasive T2 or higher urothelial cancer in past 2 years
* Participation in another clinical study involving an investigational product within 1 month before study entry
* BCG or local chemotherapy treatment (including VEGF-targeted therapy) in the upper urinary tract within 2 months prior to inclusion
* Systemic chemotherapy treatment (including VEGF-targeted therapy) within 2 months prior to enrollment
* Prohibited medication that could not be adjusted or discontinued prior to study treatment

  • Patients with photosensitive skin diseases or porphyria
* Any other medical or psychiatric co-morbidities, including decompensated heart failure, unstable angina or coronary artery disease or severe pulmonary or liver disease or current heavy smoker that, in the opinion of the study investigator, would make the patient a poor candidate for the study
* Pregnant or breast-feeding women.Women of childbearing potential (WOCBP) must undergo a negative serum pregnancy test prior to study entry.
* Men and women of reproductive potential not willing to observe conventional and effective birth control for the duration of treatment and for 90 days following the last padeliporfin VTP treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2029-01-25 (Estimated)

PRIMARY OUTCOMES:
Number of patients with absence of UTUC tumors in the entire ipsilateral calyces, renal pelvis and ureter | 28 +/- 3 days post last treatment
  Primary efficacy outcome is the absence of UTUC tumors in the entire ipsilateral calyces renal pelvis and ureter on endoscopic evaluation at the time of Primary Response Evaluation (PRE) (28 +/- 3 days post last treatment) during padeliporfin VTP induction treatment phase. This outcome will be determined dichotomously as either failure or success in achieving complete response.
  · Complete Response will be defined as absence of disease based on:
  * absence of visual tumor on endoscopy
  * no evidence of tumor on biopsy (if feasible)
  * negative urinary cytology by instrumented collection

SECONDARY OUTCOMES:
Duration of response at the entire ipsilateral kidney | 12 months post PRE
  The duration of response at the entire ipsilateral kidney will be defined as absence of disease in the entire ipsilateral calyces, renal pelvis and ureter, based on:
  * instrumented cytology
  * visually on endoscopy
  * biopsy pathology (if feasible) as will be measured at the 12 months maintenance treatment visit post PRE
Duration of response at the entire ipsilateral kidney | 3, 6, 9 months post PRE
  The duration of response at the entire ipsilateral kidney will be defined as absence of disease in the entire ipsilateral calyces, renal pelvis and ureter, based on:
  * instrumented cytology
  * visually on endoscopy
  * biopsy pathology (if feasible) as will be measured at the 3, 6, 9 months maintenance treatment visits post PRE
Duration of response at the Treatment Area of the ipsilateral kidney | 3, 6, 9, and 12 months post PRE
  Duration of response at the Treatment Area of the ipsilateral kidney will be defined as absence of disease in the ipsilateral Treatment Area, based on:
  * instrumented cytology
  * visually on endoscopy
  * biopsy pathology (if feasible) as will be measured at the 3, 6, 9, and 12 months maintenance treatment visits post PRE
Overall renal function | 6 and 12 months post PRE
  Overall renal functional outcome will be measured at the 6 and 12 months maintenance treatment visits post PRE, and will be evaluated by comparing pre-treatment and 12-month estimated glomerular filtration rate (eGFR), calculated from serum creatinine levels, using the CKD-Epi method including:
  * Absolute change in eGFR as well as categories of CKD will be utilized based on KDIGO 2012 criteria
  * Description will include change in eGFR, change in CKD stage/risk category
Kidney organ loss or preservation | 3, 6, 9, and 12 months post PRE
  Kidney organ loss or preservation will be recorded at each maintenance treatment visit post PRE at 3, 6, 9, and 12 months Maintenance Treatment visits, and will describe the reasons for organ preservation or loss. A radical nephroureterectomy, nephron-sparing surgery for UTUC or ureterectomy will be considered as organ loss.
Pathological evaluation of response | After at least one VTP treatment
  PathologicalPathological evaluation of response will be performed in kidney tissue of patients that will undergo kidney surgical removal (kidney sparing, or radical nephroureterectomy) following at least one padeliporfin VTP treatment
Patients with ureteral obstruction and/or ureteral stent | Baseline 12 months
  Patients with existing ureteral obstruction and/or existing ureteral stent will be permitted with radiographic evidence of pre-existing obstruction documented, to demonstrate the site and degree of obstruction with retrograde pyelography at baseline (prior to treatment) and will be repeated and recorded at 12 months maintenance treatment visit (post treatment) which will further be supported with CT Urogram results at 12 months to demonstrate the site and degree of obstruction using standard nomenclature.
Long Term follow-up Duration of the response | 18, 24,36,48 and 60 months post PRE or 6 and 12 months post PRE
  The duration of response in the ipsilateral kidney and treatment area will be defined as absence of disease, based on:
  * instrumented cytology
  * visually on endoscopy
  * biopsy pathology (if present and performed)
Long Term follow-up Kidney organ loss or preservation | 18, 24,36,48 and 60 months post PRE or 6 and 12 months post PRE
  Kidney organ loss or preservation will be recorded and will describe the reasons for organ preservation or loss. A radical nephroureterectomy, nephron-sparing surgery for UTUC or ureterectomy will be considered as organ loss and a pathology report of the removed tissue will be recorded (if available or feasible)
Long Term follow-up Overall renal functional | 18, 24,36,48 and 60 months post PRE or 6 and 12 months post PRE
  Overall renal functional outcome will be evaluated by estimated glomerular filtration rate(eGFR) using CKD-Epimethod
Long Term follow-up Safety Follow up | 18, 24,36,48 and 60 months post PRE or 6 and 12 months post PRE
  Safety follow up based and recording of adverse events
Exploratory Endpoint | Baseline
  Blood,tumor and cytology samples will be collected, centrally stored and later submitted for tumor genomic sequencing studies to explore the tumor genomic alterations, and mutation status as biomarkers with association to treatment response and progression events such as recurrence, grade transformation, increased stage and metastases.
Pharmacokinetic Endpoint Cmax | 0 (before injection) and 20, 40, 60, 90, 120 and 360 mn after end of injection
  Patients with moderate hepatic impairment, will undergo a pharmacokinetic evaluation, blood samples will be collected to evaluate Cmax
Pharmacokinetic Endpoint Tmax | 0 (before injection) and 20, 40, 60, 90, 120 and 360 mn after end of injection
  Patients with moderate hepatic impairment, will undergo a pharmacokinetic evaluation, blood samples will be collected to evaluate Tmax
Pharmacokinetic Endpoint T1/2 | 0 (before injection) and 20, 40, 60, 90, 120 and 360 mn after end of injection
  Patients with moderate hepatic impairment, will undergo a pharmacokinetic evaluation, blood samples will be collected to evaluate T1/2
Pharmacokinetic Endpoint AUC | 0 (before injection) and 20, 40, 60, 90, 120 and 360 mn after end of injection
  Patients with moderate hepatic impairment, will undergo a pharmacokinetic evaluation, blood samples will be collected to evaluate AUC
Pharmacokinetic Endpoint CL | 0 (before injection) and 20, 40, 60, 90, 120 and 360 mn after end of injection
  Patients with moderate hepatic impairment, will undergo a pharmacokinetic evaluation, blood samples will be collected to evaluate CL

CONTACTS AND LOCATIONS:
Overall Officials: Vitaly Margulis, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (18):
- United States (12):
  - University of California - Irvine Medical Center, Irvine, California
  - Keck School of Medicine at USC Medical Center, Los Angeles, California
  - Emory University Hospital, Atlanta, Georgia
  - The Johns Hopkins Hospital, The Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Albany Medical College, Albany, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Ohio State University (OSU), Columbus, Ohio
  - The Pennsylvania State University (Penn State) Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - University of Texas Southwestern, Dallas, Texas
  - University of Washington, Seattle, Washington
- France (2):
  - CHU de Lille - Hopital Claude Huriez, Lille
  - HCL Hopital Edouard Herriot, Lyon
- Universitaetsklinikum Tuebingen, Tübingen, Germany
- Sheba Medical Center, Ramat Gan, Israel
- Spain (2):
  - Hospital Universitario de A Coruña, A Coruña
  - Hospital Universitario Vall d'Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: No